CLINICAL TRIAL: NCT04348669
Title: Tele-yoga and Dystonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jean-Francois Daneault, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020000758
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Cervical Dystonia
Keywords: yoga; cervical dystonia; telerehabilitation
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Intervention Model Description: This is a single group intervention study of adults (18-80 years-old) with cervical dystonia undergoing a 6-week intervention of 30-minute yoga classes delivered remotely through videoconferencing 2 times per week. There will be baseline testing (0-weeks), post-intervention testing (6-weeks), and follow-up testing (12-weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-yoga (Experimental): This is a single group study with all subjects included in this single arm. All subjects will undergo the same telerehabilitation yoga intervention delivered through videoconferencing.
  Interventions: Other: Tele-yoga

INTERVENTIONS:
Other: Tele-yoga — Subjects will undergo 30-minute yoga sessions delivered remotely 2 times/week for 6-weeks. The yoga sessions will be delivered one-on-one. The sessions will include 5-7 minutes of breathing exercises, 15-20 minutes of postures, and 5-7 minutes of relaxation and meditation exercises.

SUMMARY:
The purpose of this study is to investigate the effect of yoga delivered remotely on adults with dystonia. This work will have implications related to physical interventions symptom management and quality of life as well as implications related to the role of tele-therapy.

DETAILED DESCRIPTION:
This is a single group intervention study of adults (18-80 years-old) with dystonia symptoms undergoing a 6-week intervention of 30 minute yoga classes delivered remotely through videoconferencing 2-3 times a week. Subjects with cervical dystonia will complete yoga classes delivered at-home with videoconferencing, receiving one-on-one yoga instruction including breathing, postures, and meditation/relaxation for two to three times a week. Data collection will occur remotely via videoconferencing at 0-weeks (baseline), 6-weeks (after the intervention), and 12-weeks (follow-up). Data collection will include demographics, mental health questionnaires, motor assessments, enjoyment, usability, and follow-up yoga status. Each yoga session will be video recorded to aide in recording adherence, adverse events, and challenges.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of cervical dystonia
2. 18-80 years old
3. Ability to communicate verbally and follow directions
4. English-Speaking
5. Subject has access to WiFi and applicable technological device (computer, laptop, tablet, smartphone etc)
6. Subject is willing to be video recorded during the yoga session
7. Subject is willing to open Zoom on their technological device
8. Subject feels comfortable using a technological device for the intervention (ie demonstrates self-reported technological literacy)

8) if they are a U.S. resident, they must be a New Jersey resident and will participate in a majority of the intervention sessions from New Jersey. International enrollment will be considered on a case-by-case basis based on the Physical Therapy Licensure regulations of the appropriate Physical Therapy board.

Exclusion Criteria:

1. Diagnosis of major depressive disorder,
2. Injury or condition that could prevent the ability to engage in yoga poses based on self-report
3. Cognitive impairment or condition that would prevent the subject from understanding the tasks or communicating with the research team
4. Past yoga experience exceeding 5 or more times within the last 2 months
5. pregnant women
6. No access to a technological device (such as a smartphone, computer, laptop, or tablet) or access to WiFi that can be used to access the teleconferencing medium
7. If the subject does not want to be recorded during the yoga sessions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Craniocervical Dystonia Questionnaire (CDQ-24) | Baseline (0-weeks)
  The 24-question CDQ-24 will be used to measure disease-specific quality of life. It is comprised of five categories, which are stigma, emotional well-being, pain, activities of daily living (ADL), and social and family life. Potential scores range from 0-100 with higher scores indicating worse quality of life.
Craniocervical Dystonia Questionnaire (CDQ-24) | Post-intervention (6-weeks)
  The 24-question CDQ-24 will be used to measure disease-specific quality of life. It is comprised of five categories, which are stigma, emotional well-being, pain, activities of daily living (ADL), and social and family life. Potential scores range from 0-100 with higher scores indicating worse quality of life.
Craniocervical Dystonia Questionnaire (CDQ-24) | Follow-up (12-weeks)
  The 24-question CDQ-24 will be used to measure disease-specific quality of life. It is comprised of five categories, which are stigma, emotional well-being, pain, activities of daily living (ADL), and social and family life. Potential scores range from 0-100 with higher scores indicating worse quality of life.

SECONDARY OUTCOMES:
Short form 36 health survey (SF-36) | Baseline (0-weeks), post-intervention (6-weeks) and at follow-up (12-weeks)
  The SF-36 will be used to assess quality of life. It is a 36-item questionnaire that consists of eight domains: physical functioning (PF), role limitations due to physical health (RP), role limitations due to emotional problems (RE), vitality (VT), mental health, social functioning (SF), bodily pain (BP), and general health (GH). With higher scores indicating greater quality of life.
Beck Anxiety Scale (BAI) | Baseline (0-weeks), post-intervention (6-weeks) and at follow-up (12-weeks)
  The BAI will be used to measure symptoms of anxiety. The BAI is a brief measure of anxiety with a focus on somatic symptoms of anxiety. Respondents indicate how much they have been bothered by each symptom over the past week. Responses are rated on a 4-point Likert scale and range from 0 (not at all) to 3 (severely). Potential scores range from 0 to 63 with higher scores indicating greater symptoms of anxiety.
Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) | Baseline (0-weeks), post-intervention (6-weeks) and at follow-up (12-weeks)
  The TWSTRS- severity scale will be used to assess motor symptoms. The TWSTRS is a comprehensive scale designed to assess objective physical (severity subscale) and subjective findings (disability and pain subscales). With higher scores indicating greater severity of symptoms.
Beck Depression Inventory-II (BDI-II) | Baseline (0-weeks), post-intervention (6-weeks) and at follow-up (12-weeks)
  BDI-II will be used to measure symptoms of depression. The BDI-II is a 21 item self-report measure. For each item the subject must choose one out of 4 statements of increasing severity regarding a specific symptom of depression. It is written approximately at a 5th grade reading level and takes about 5-10 minutes to complete. Potential scores range from 0-63 with higher scores indicating greater severity of depressive symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Baseline (0-weeks), post-intervention (6-weeks) and at follow-up (12-weeks)
  The PSQI will be used to assess sleep dysfunction. The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Potential scores range from 0-21 with higher scores indicating greater sleep dysfunction.
Five Times Sit to Stand Test (FTST) | Baseline (0-weeks), post-intervention (6-weeks) and at follow-up (12-weeks)
  The FTST, functional measure, will be administered to assess physical function. It will be administered using a chair in the participants' homes over a one-on-one Zoom videoconference. Participants will be encouraged to have another adult present during this portion of the data collection in case there is any loss of balance. Participants will be encouraged to use an armless chair approximately 63 centimeters from the ground and any deviation from this standard procedure will be documented. Time in seconds it takes the participant to raise from the chair 5 times will be recorded. Longer times will indicate poorer physical function.
Adherence will be assessed by calculating the total number of yoga sessions attended. | Between week 0 to week 6
  Adherence to the yoga classes will be recorded each class including if a class is rescheduled. The occurrence, frequency, and brief description of any home yoga practice will also be recorded.
Adverse Events | Between week 0 to week 6
  All adverse events will be documented with a brief description of each adverse event, the potential relationship to the study, and the severity of each event.
Technical Difficulties Encountered | Between week 0 to week 6
  Anything perceived has a challenge by the yoga instructor or participant will be will be documented with severity of the challenge measured by time disrupted at an event level (time disrupted by the single event) and time disrupted from an entire session (time disrupted cumulatively).
Enjoyment/Feedback | Post-intervention testing (at 6-weeks)
  Enjoyment/feedback will be assessed via a Qualtrics questionnaire created by the study team inquiring about the subject's opinions about the intervention and a 10-point enjoyment scale.
Usability | Post-intervention testing (at 6-weeks)
  The systems usability scale, a 10-item scale that will be used to assess how usable the subjects feel that the tele-yoga intervention was. Scores are calculated such that a total score of 100 is possible. Higher scores indicate higher usability.
Yoga Status at Follow-up | Follow-up (12 weeks)
  Yoga status at follow-up will be assessed via a Qualtrics questionnaire created by the study team asking questions about the subject's current involvement in yoga and other related topics.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Daneault, Principal Investigator — Rutgers University
Locations (1):
- Motor Behavior Laboratory, Newark, New Jersey, United States